CLINICAL TRIAL: NCT02567721
Title: European Medicines Agency (EMA) Post-authorisation Safety Study of Influenza Vaccine
Brief Title: Post-authorisation Safety Study (PASS) of Influenza Vaccine in United Kingdom (UK)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 202055
Record Dates: First submitted 2015-09-18; First posted 2015-10-05 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Influenza
Keywords: Post-authorisation safety study (PASS); Adverse Drug Reaction Reporting Systems; Post marketing product surveillance; European Medicines Agency (EMA); Influenza Vaccine; Computerized Medical Record System; United Kingdom; Primary Health Care
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

GROUPS / COHORTS (1):
- Study Cohort: Subjects who will receive influenza vaccination between 1 September 2015 and 30 November 2015 in the 9 GP practices from who clinical data routinely collected as part of clinical consultations in primary care will be extracted.
  Interventions: Other: Vaccine safety surveillance

INTERVENTIONS:
Other: Vaccine safety surveillance — Extraction of routinely collected primary care data from nine GP practices and an active surveillance approach in 3 of the 9 GP practices, by using an existing card-based ADR reporting system (MHRA Yellow Card), to estimate proportions of AEIs among seasonal influenza-vaccinated individuals.
  Other Names: Data collection

SUMMARY:
The purpose of this study is to conduct a pilot study to explore the potential use of routinely collected data in General Practitioner (GP) practices to conduct enhanced safety surveillance of seasonal influenza vaccines in the UK, as recommended in the EMA interim guidance on enhanced safety surveillance for seasonal influenza vaccines in the EU.

DETAILED DESCRIPTION:
Data routinely collected as part of clinical consultations in primary care will be extracted from nine General Practitioner (GP) practices in order to estimate medically attended Adverse Events of Interest (AEIs), for people who have received an influenza vaccine. This study will also actively follow patients who were exposed to seasonal influenza vaccination for 7 days in three of the nine GP practices using a customised card-based adverse drug reaction reporting system, in order to determine whether a more active approach to surveillance can capture higher rates of AEIs.

ELIGIBILITY:
Inclusion Criteria:

* All individuals (aged 6 months and above) who will receive seasonal influenza vaccination in the 9 GP practices between 1 September 2015 and 30 November 2015.
* Pregnant women are also included in this study.

Exclusion Criteria:

• Only registered patients who have explicitly opted out of data sharing will be excluded from the analysis.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Registered patients in 9 GP practices in England and who are immunized against seasonal influenza between 1 September 2015 and 30 November 2015
Sampling Method: Non-Probability Sample
Enrollment: 11530 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of patient counts of the total registered patients vaccinated by age strata, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
Proportions of total registered patients vaccinated by age strata, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
Number of patient counts of the total registered patients vaccinated by co-morbidity, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
Proportions of total registered patients vaccinated by co-morbidity, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
Number of patient counts of the vaccinated patients with reported endpoints of interest by age strata, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
  - Presentation with fever or other febrile illness, - Presentation related to local reaction, - Presentation related to general reaction (fatigue, myalgia, etc.), - All other presentations that could plausibly be related to vaccination.
Proportions of vaccinated patients with reported endpoints of interest by age strata, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
  - Presentation with fever or other febrile illness, - Presentation related to local reaction, - Presentation related to general reaction (fatigue, myalgia, etc.), - All other presentations that could plausibly be related to vaccination.
Number of patient counts of the vaccinated patients with reported endpoints of interest by co-morbidity, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
  - Presentation with fever or other febrile illness, - Presentation related to local reaction, - Presentation related to general reaction (fatigue, myalgia, etc.), - All other presentations that could plausibly be related to vaccination.
Proportions of vaccinated patients with reported endpoints of interest by co-morbidity, reported weekly and cumulatively by brand (also indicating those for whom brand data are unavailable) | Up to 3 months (between 1 September 2015 and 30 November 2015)
  - Presentation with fever or other febrile illness, - Presentation related to local reaction, - Presentation related to general reaction (fatigue, myalgia, etc.), - All other presentations that could plausibly be related to vaccination.

SECONDARY OUTCOMES:
Completeness of vaccination data in the computerized medical record system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Completeness of AEI reporting in the computerized medical record system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Timeliness of vaccination data in the computerized medical record system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Timeliness of AEI reporting in the computerized medical record system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Completeness of vaccination data in the card-based adverse event reporting system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Completeness of AEI reporting in the card-based adverse event reporting system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Timeliness of vaccination data in the card-based adverse event reporting system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Timeliness of AEI reporting in the card-based adverse event reporting system. | Up to 3 months (between 1 September 2015 and 30 November 2015)
Incidence rates for the 5 most frequently reported AEs reported alongside those available in the literature from a similar population (vaccinated or general population if vaccinated not available) within the same risk period and stratified by age. | Up to 3 months (between 1 September 2015 and 30 November 2015)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Surrey, United Kingdom